CLINICAL TRIAL: NCT05030597
Title: Exploring the Application Value of PET Molecular Imaging Targeting FAP in Oral Squamous Cell Carcinoma
Acronym: FAPI-OSCC
Status: Recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PTXM2021021
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-07

CONDITIONS: PET/CT; FAPI; Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Gallium-68; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 68Ga-DOTA-FAPI and 18F-FDG PET/CT: Investigators recruit patients whom are clinically highly suspected oral cancer or recurrence after treatment. Patients undergo baseline 68Ga-FAPI and 18F-FDG PET/CTwithin one week. For resectable locally advanced cases receiving neoadjuvant therapy from oral and maxillofacial clinicians, a follow-up FAPI PET imaging will be performed after two cycles of treatment and before surgery.
  Interventions: Drug: 68Ga-DOTA-FAPI; Device: PET/CT; Diagnostic Test: Participants receive baseline paired FDG and FAPI PET/CT. For resectable locally advanced cases receiving neoadjuvant therapy undergo follow-up FAPI PET imaging.

INTERVENTIONS:
Drug: 68Ga-DOTA-FAPI — Intravenous access is pre-established. Quality control is carried out to confirm the radiochemical purity of 68Ga-DOTA-FAPI by HPLC. Intravenous administration of 68Ga-DOTA-FAPI according to 1.85-3.7 MBq/kg body weight (0.05-0.1 mCi/kg), rinsed with 0.9% saline, and hydrated after drinking more water.
  Other Names: gallium-68 (68Ga)-Fibroblast activation protein inhibitor (FAPI)
Device: PET/CT — Each subject undergoes PET/CT imaging within 20-30 minutes after injection.
  Other Names: Positron Emission Tomography/Computed Tomography
Diagnostic Test: Participants receive baseline paired FDG and FAPI PET/CT. For resectable locally advanced cases receiving neoadjuvant therapy undergo follow-up FAPI PET imaging. — This observational study evaluates the application of paired FDG and FAPI PET/CT in oral cancer.
  1. Baseline phase: All participants undergo baseline FDG and FAPI PET/CT scans.
  2. Post-neoadjuvant phase: For patients with resectable locally advanced disease receiving neoadjuvant therapy (as per clinician decision), a second FAPI PET/CT scan is performed after 2 cycles of treatment to assess treatment response.
  3. Purpose: To explore the utility of FAPI PET in (a) initial staging, (b) treatment response evaluation, and (c) prognostic value in oral cancer.

SUMMARY:
In this prospective study, the investigators will use integrated PET/CT with the agent 68Ga-FAPI and conventional imaging agent 18F-FDG to explore the application value of FAP-targeted molecular imaging in the diagnosis and staging for oral cancer. This study also aims to explore the application value of FAPI imaging in evaluating treatment response for oral cancer.

DETAILED DESCRIPTION:
Positron emission tomography (PET) molecular imaging provides a valuable method for the diagnosis, differential diagnosis and staging of various tumors. Cancer associated fibroblasts (CAFs) are the main components of tumor stroma, which are involved in tumor cell proliferation, invasion, metastasis and tumor angiogenesis, and play an important role in the occurrence and development of tumors. Fibroblast activation protein (FAP) is the most potential specific molecular marker of CAF, which is mainly expressed in stromal fibroblasts of epithelial tumors and is a potential molecular target for tumor diagnosis and treatment. Oral cancer is the most common type of malignant head and neck cancer, seriously endangering human health. Accurate delineation of the primary tumor, detection of regional nodal metastases, distant metastases and second primary tumors are important for determining the therapeutic strategy and prognosis of oral cancer. Currently, the molecular imaging agent most commonly used in clinical practice for oral cancer is 18F-fluoro-deoxy-glucose (18F-FDG). However, 18F-FDG exhibits some shortages. Inflammatory lesions and the surrounding normal tissue such as brain, tonsils and salivary glands show high uptake of 18F-FDG, often affecting the judgment of lesions.

Adult patients aged >18 years with clinically confirmed or highly suspected oral cancer will be enrolled. Participants receive paired baseline FDG and FAPI PET/CT to explore the diagnostic and staging value of FAPI PET in oral cancer. For resectable locally advanced cases receiving neoadjuvant therapy from oral and maxillofacial clinicians, a follow-up FAPI PET imaging will be performed after two cycles of treatment and before surgery to evaluate its application in treatment-response assessment. Ultimately, this study aims to comprehensively evaluate the clinical utility of FAPI PET/CT in oral cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent;
2. Aged 18~70 years;
3. Clinically highly suspected oral cancer and recurrence after treatment (Newly diagnosed patients: Scheduled for surgery or neoadjuvant therapy followed by surgery);
4. Ability to complete baseline and follow-up PET/CT (Follow-up FAPI PET/CT applies only to locally advanced patients undergoing neoadjuvant therapy.).

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning pregnancy during the trial period;
2. Known hypersensitivity to FAPI, FDG, or their components, or history of severe allergic reactions;
3. People with poor general condition, their heart, lung, liver, kidney and other important organ functions cannot tolerate surgery;
4. Before the injection of 18F-FDG, the fasting blood glucose level exceeded 11.0 mmol/L;
5. Claustrophobia or inability to tolerate PET/CT imaging (Those who cannot tolerate lying supine for 15~30 minutes.);
6. Participation in another interventional clinical trial within 30 days prior to enrollment, or planned participation during this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls adults aged 18-70 years with clinically suspected or histopathologically confirmed oral cancer (primary or recurrent). Newly diagnosed patients are scheduled for surgery or neoadjuvant therapy, while recurrent cases require imaging/pathology confirmation. All participants must complete baseline FAPI PET/CT and FDG PET/CT for diagnostic/staging evaluation. Locally advanced patients receiving neoadjuvant therapy will undergo follow-up FAPI PET/CT for therapeutic response assessment. Exclusion criteria include pregnancy, severe allergies to FAPI/FDG, uncontrolled comorbidities, and recent participation in other interventional trials.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance (sensitivity, specificity, accuracy) and staging of FAPI PET in oral cancer | Baseline (at initial diagnosis, prior to treatment)
  Comparison of FAPI PET and FDG PET in diagnosing oral cancer, including sensitivity, specificity, accuracy, and TNM staging. Assessments performed at baseline using histopathology and imaging as reference standards.

SECONDARY OUTCOMES:
FAPI PET for therapeutic response evaluation | After completion of 2nd cycle of neoadjuvant therapy, just prior to surgery
  Assessment of FAPI PET parameters for predicting treatment response in patients receiving neoadjuvant therapy. Follow-up FAPI PET performed post-treatment.
Prognostic value of FAPI PET parameters in oral cancer | Through study completion, an average of 1 year
  Correlation between FAPI PET parameters and long-term outcomes (e.g., progression-free survival, overall survival).
Correlation between FAPI PET parameters and histopathological biomarkers | At baseline and 6 weeks post-FAPI PET scan
  Correlation between FAPI PET parameters (SUVmax/SUVmean/SUVpeak) and histopathological biomarkers of tumor tissue.
  1. FAP expression level (H-score; immunohistochemistry)
  2. PD-L1 expression (Combined Positive Score; Dako 22C3 IHC assay)
  3. CD8 expression (H-score; immunohistochemistry)
  4. Granzyme B expression (H-score; immunohistochemistry)

CONTACTS AND LOCATIONS:
Overall Officials: He Yong, PhD, Study Chair — Zhongnan Hospital
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzgerald AA, Weiner LM. The role of fibroblast activation protein in health and malignancy. Cancer Metastasis Rev. 2020 Sep;39(3):783-803. doi: 10.1007/s10555-020-09909-3. PMID 32601975
- [Background] Syed M, Flechsig P, Liermann J, Windisch P, Staudinger F, Akbaba S, Koerber SA, Freudlsperger C, Plinkert PK, Debus J, Giesel F, Haberkorn U, Adeberg S. Fibroblast activation protein inhibitor (FAPI) PET for diagnostics and advanced targeted radiotherapy in head and neck cancers. Eur J Nucl Med Mol Imaging. 2020 Nov;47(12):2836-2845. doi: 10.1007/s00259-020-04859-y. Epub 2020 May 23. PMID 32447444
- [Background] Chen H, Pang Y, Wu J, Zhao L, Hao B, Wu J, Wei J, Wu S, Zhao L, Luo Z, Lin X, Xie C, Sun L, Lin Q, Wu H. Comparison of [68Ga]Ga-DOTA-FAPI-04 and [18F] FDG PET/CT for the diagnosis of primary and metastatic lesions in patients with various types of cancer. Eur J Nucl Med Mol Imaging. 2020 Jul;47(8):1820-1832. doi: 10.1007/s00259-020-04769-z. Epub 2020 Mar 28. PMID 32222810
- [Derived] Jiang Y, Yu Z, Sun Y, Tian Y, Wang L, Xing D, Huang Y, He Y, Jia J. Predictive value of [68Ga]Ga-FAPI-04 PET/CT on pathologic response to neoadjuvant chemoimmunotherapy for locally advanced resectable oral squamous cell carcinoma. Eur J Nucl Med Mol Imaging. 2025 Dec;53(1):283-294. doi: 10.1007/s00259-025-07414-9. Epub 2025 Jun 23. PMID 40548990